CLINICAL TRIAL: NCT06817304
Title: Tiny Heroes: Decrease and Prevent Anxiety Problems in Young Children - a Feasibility Study
Brief Title: Tiny Heroes: Decrease and Prevent Anxiety Problems in Young Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Lalouni, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-07258-01
Record Dates: First submitted 2025-01-21; First posted 2025-02-10 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Anxiety, Mild to Moderate; Inhibited Temperament
Keywords: preschool anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is a behavioral intervention, therefore study phase is not applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent-directed online cognitive behavioral therapy (Experimental)
  Interventions: Behavioral: Tiny Heroes

INTERVENTIONS:
Behavioral: Tiny Heroes — This is a four modules online intervention based on cognitive behavioral therapy directed at parets of anxious children 3-6 years

SUMMARY:
In Sweden, there is a lack of evidence-based methods to reduce and prevent young children's emotional problems, such as worry and anxiety. In the project, the intervention Tiny Heroes will be evaluated in an open feasibility trial.

Tiny Heroes is an online cognitive behavioral therapy (iCBT) directed at parents, adapted to the Swedish clinical setting in workshops with clinicians and health care developers in Region Stockholm. Feedback from parents will be included in the feasibility study and inform the intervention.

Research questions

* Is Tiny Heroes preliminary effective in reducing children's anxiety symptoms?
* What support is needed from clinicians during Tiny Heroes?
* How many modules are completed by parents?
* How is Tiny Heroes perceived by parents?

If Tiny Heroes is feasible and preliminary effective, a randomized controlled trial will be planned for (not included in this project plan).

DETAILED DESCRIPTION:
Anxiety is the most prevalent mental disorder in children and the most commonly reported reason for children having contact with first-line mental healthcare. In pre-school children, the most prevalent anxiety disorders are specific phobia (i.e., exaggerated fear in specific situations or of certain objects), social anxiety (i.e., fear in social situations), and separation anxiety (i.e., fear of being separated from parents or other significant persons). Childhood anxiety may impact many areas of the child's functioning, including the family, preschool, and peer relations. It is predictive of anxiety, depression and substance abuse in later childhood and adulthood. Due to this over-time comorbidity, there has been a move towards developing interventions for very young children.

Behavioral inhibition is a temperamental trait associated with anxiety in children. Behavioral inhibition is characterised by avoidance behaviors, behaviours aiming to maintain proximity to safety figures, distress when dealing with novelty, and socially withdrawn behaviors. A parenting style that has been associated with childhood anxiety is overprotective parenting. Parents are the most important and influential persons for young children. If parents receive appropriate support, they can positively influence how their child learn to deal with difficult emotions and situations. According to the transactional model, anxiety in childhood develops from the interplay between child temperament and parenting. A child who is high in behavioral inhibition will elicit overprotective parenting, which in turn will reinforce inhibited and withdrawn behaviours. In CBT, this vicious circle is targeted by trying to decrease both overprotective parenting and the child's behavioral avoidance.

CBT is the first-line treatment for anxiety in children, but very few young children receive CBT. A recent Cochrane analysis recommends research about how to make CBT more accessible and how to reach neglected populations. Internet platforms, such as the national platform Stöd och behandling, offer a possibility to scale up CBT and thereby making it available to more families. Online CBT directed at parents has recently been found to be non-inferior to treatment as usual in a large randomized controlled trial for anxiety in young children. Because less resources are needed when administering online treatments compared to face-to-face treatments, resources can then be unlocked for families with pressing needs. Families can engage in online interventions without taking time off from work and engage in the intervention at a time that fit their lives. The content is structured and thereby quality assured, and it can easily be translated to different languages, enabling parents who don't comprehend Swedish to take part of the treatment.

In Sweden, first-line mental healthcare units are commissioned to help children with mild to moderate anxiety. For the youngest children (0-5 years) in Region Stockholm, six MALINA clinics offer these services. The clinicians at MALINA are psychologists and the level of care lies between child health services (BVC) and child and adolescent mental health services (BUP). The standard treatment for children with anxiety problems at MALINA today is information to parents about anxiety and how they can support their anxious children.

Most mental health interventions are developed for the use in a mental health care setting and very few protocols have been fitted to first-line mental healthcare clinics. Interventions in first-line mental healthcare are generally shorter and oftentimes clinicians make ad-hoc adjustments in which they shorten interventions. Thus, interventions are often provided in a way that differ distinctively from how they were evaluated.

The present project will fill important gaps in clinical practice and research by co-developing and fitting cognitive behavioral therapy (Tiny Heroes) for young children with mild to moderate anxiety problems to first-line mental healthcare at MALINA.

The purpose of targeting parents of young children is twofold: First, it enables children to be offered support via their most influential persons - their parents. Second, the parents will be able to give continuous support to their children over many years, which may enable prevention of future anxiety. Even though parental support is recommended for young children with anxiety, such programs are lacking in Swedish healthcare today, which is why Tiny Heroes will fill an important gap in treatment and research.

The project is a collaboration between Center for Epidemiology and Community Medicine (CES) in Region Stockholm, MALINA (all six MALINA units in Region Stockholm will be involved), Karolinska Institutet, and the Child Health Care unit in Region Stockholm (which supports MALINA via healthcare developers). The families will receive Tiny Heroes as part of their health care at MALINA. However, the data collection: online questionnaires, clinical assessments, and a qualitative workshop after the intervention will be conducted by Karolinska Institutet

In the present study, caretakers/parents of 20 children will be recruited to the study at MALINA. If there are two (or more) caretakers/parents, only one will be asked to participate in the study (but both caretakers/parents are expected to take part in the Tiny Heroes intervention). Psychologists at MALINA will check the inclusion and exclusion criteria. Eligible parents interested in participating in the study, will use a link provided by MALINA to the secure internet platform REDCap were informed consent will be collected and questionnaires will be assessed.

All questionnaires will be self-assessed by the parents within the web application Research Electronic Data Capture (REDCap), provided by Karolinska Institutet. Assessments will be collected at baseline, at follow-up after the intervention six weeks after baseline, and at follow-up assessment 3 months after the end of the intervention. ADIS-P will be assessed in a digital clinical interview with the parent using a closed meeting in the KI Zoom platform. The interview will be recorded, and the audio file will be saved on a secure and encrypted server space at KI. The audio files will be stored until the manuscript from the study is published, to enable quality checks. After that, it will be deleted.

After each module, parent will be asked to provide short written feedback about the module by answering questions about the modules content and its technical function.

All parents who participate in the program and who consent to be asked about participating in a workshop at the end of the program will be invited to participate in such a workshop after the Tiny Heroes program. Participation is voluntary. The workshop will use adaptive reflection, in which parents first reflect individually, then together in the group, on different aspects of the Tiny Heroes intervention. The feedback will be transcribed during the workshop and the written material will be saved on a secure server at Karolinska Institutet.

Assessments will be conducted at baseline, at follow-up after the intervention, and at follow up assessment 3 months after the intervention. The preliminary effects will be evaluated using dependent t-tests, comparing the mean levels of the measures between baseline and after treatment, between assessments after treatment and three months follow-up, and between assessment at baseline and three months follow-up. Cohen's d effect sizes will be based on the standardized mean differences between the assessments at these time points. Results on the Client satisfaction questionnaire and Adverse Events scale will be presented with descriptive statistics. Power was based on attaining a moderate within-group effect size (d= 0.69) on PAS found in a previous similar study and gives an 80% power to detect differences with an alpha level of .05, also accounting for 15% dropouts.

The written feedback from the parents (attained after each module) and the feedback from the workshop with the parents will be analyzed using thematic analysis. The output will be used to inform possible changes to the Tiny Heroes intervention.

The present study may fill important gaps in both clinic and research because there is a lack of evidence-based interventions for young children with mild to moderate anxiety problems within first-line mental healthcare. Today, many children with anxiety problems don't receive adequate help. Even though CBT with significant parental involvement is recommended for the treatment of anxiety in young children, there is a lack of such methods. Digital interventions directed at parents have been highlighted as a way to increase the number of children treated for anxiety problems without compromising treatment outcomes. An intervention similar to Tiny Heroes was recently found effective and also credible by parents and therapists. Another feature that contributes to the quality of the study is that co-development was used in the development of Tiny Heroes.

Most evidence-based methods are not developed within the same setting as they used. Here, clinicians from MALINA, have been involved from the start. Discussions about the length, type of treatment, delivery format, treatment components, and adjustments to fit the intervention into regular care informed the development of Tiny Heroes. During 2023, the research group preliminary tested the treatment Cool Little Kids, also targeting parents of anxious children aged 3-6 years. Group discussions with the parents included in this testing informed the decision to instead develop the online program Tiny Heroes. Among other things, the parents expressed a need of making the treatment more accessible and possible to take part of outside office hours, hence the online format.

Tiny Heroes may fill an important treatment gap by offering an structured early intervention for very young children with anxiety problems. The parent-based intervention will be offered at a time in the children's lives, when parents are very influential. In Tiny Heroes, parents encourage their children to increase brave behaviors and to decrease avoidant behaviors, in a step-by-step manner. This will likely help children engage in more activities in their daily lives. It may shift children's future trajectories from anxious and avoidant paths to more active and healthy ones.

The internet format of Tiny Heroes offers a unique opportunity to ensure that families get exactly the treatment evaluated in research. If proven effective, access to Tiny Heroes can easily be scaled up and translated to commonly used languages in Sweden. Thus, it has the capacity to increase access to evidence-based interventions in the community and decrease inequalities in health.

ELIGIBILITY:
Inclusion criteria:

* Parent or caretaker of child 3-6 years with primary problem of worries, fear, or anxiety, assessed by a licensed psychologist at MALINA
* Parent or caretaker can read Swedish
* Parent or caretaker has access to computer, tablet or mobile phone with internet connection

Exclusion criteria:

* Child having major developmental disorder (e.g., intellectual disability or severe autism spectrum disorder)
* Parent having significant intellectual impairment or mental health problems (likely to interfere with participation in the treatment)
* Social problems which the psychologist at MALINA appraise will hinder participation in Tiny Heroes (e.g., ongoing separation between parents, serious problems with the child's pre-school)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The clinical severity rating (CSR) of ADIS-P | From enrollment to follow up at 3 months after treatment completion.
  Clinical diagnostic status will be determined with Anxiety Disorders Interview Schedule for DSM-V: Parent version (ADIS-P), pre treatment, post treatment and 3 months post treatment

SECONDARY OUTCOMES:
Preschool Anxiety Scale | From enrollment to follow up at 3 months after treatment completion.
  Child anxiety will be assessed with the Preschool Anxiety Scale. The PAS is a 34-item measure assessed by parents, pre treatment, post treatment and 3 month post treatment. Subscales align with the DSM-V anxiety diagnoses. The PAS has shown moderate to good psychometric properties with good internal consistency.
Brief Parental Self-Efficacy Scale (BPSES). | From enrollment to follow up at 3 months after treatment completion.
  Parental self-efficacy will assessed with the Brief Parental Self-Efficacy Scale (BPSES). BPSES is a five item scale that has shown a satisfactory level of internal consistency (Cronbach's alpha 0.75) . It was originally developed for the use in parents with children who displayed disruptive behavior. The research group has translated the scale to Swedish and adapted it to fit parents whose children suffer from anxiety. Parents included in the study will fill out the scale pre, post and 3 months post treatment.
Family Accommodation Scale Anxiety (FASA) | From enrollment to follow up at 3 months after treatment completion.
  Family accommodation to the child's anxiety is assessed with Family Accommodation Scale Anxiety (FASA). The scale consists of 13 items about how the family accommodates to the child's anxiety. It has shown good internal consistency and also convergent and divergent validity. Parents will fill out the questionnaire. Pre, post and 3 months post treatment.
Child Anxiety Life Interference Scale - Preschool version (CALIS-PV). | From enrollment to follow up at 3 months after treatment completion.
  Life interference will be assessed with the Child Anxiety Life Interference Scale - Preschool version (CALIS-PV). CALIS-PV is an 18-item parent-assessed scale assessing interference of child's anxiety on the child's life and the life of the parent. It has shown good validity and internal consistency. Parents will fill out the questionnaire pre, post and 3 months post treatment.

OTHER OUTCOMES:
Client satisfaction questionnaire (CSQ-8) | Assessed only once at follow-up six weeks after the baseline assessment.
  Treatment satisfaction will be assessed by the parents with the 8-item questionnaire the Client satisfaction questionnaire (CSQ-8)
Adverse Events scale (AE) | Assessed only once at follow-up six weeks after the baseline assessment.
  Negative effects of the intervention will be assessed with the Adverse Events scale (AE).
Written feedback from parents | From enrollment to end of treatment (4-6 weeks depending on speed of treatment progression)
  After each module, parent will be asked to provide short written feedback about the module by answering questions about the modules content and its technical function.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Stockholm, Karolinska Institutet
  - Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: No
This has not been included in the consent form to the participants.